CLINICAL TRIAL: NCT02674022
Title: Screening for Metabolic Problems in Women, and Possible Treatment With Vitamin/Mineral Supplement
Brief Title: Screening for Metabolic Problems in Mothers of Children With Autism and Typically Developing Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Bryan K. Woodruff, Assistant Professor of Neurology, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-006909
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy; Autistic Disorder; Folic Acid Deficiency
Keywords: Maternal Health; Autistic Disorder; Metabolism; Folic Acid
MeSH Terms: conditions — Autistic Disorder; Folic Acid Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mothers of Children with ASD (Active Comparator): Initial treatment with standard prenatal supplement in mothers with abnormal homocysteine levels; additional treatment with optimized prenatal supplement in mothers not responding adequately to initial treatment.
  Interventions: Dietary Supplement: Prenatal supplement
- Mothers of Typically Developing Children (Active Comparator): Initial treatment with standard prenatal supplement in mothers with abnormal homocysteine levels; additional treatment with optimized prenatal supplement in mothers not responding adequately to initial treatment.
  Interventions: Dietary Supplement: Prenatal supplement

INTERVENTIONS:
Dietary Supplement: Prenatal supplement — Treatment with a standard and optimized prenatal supplement, dependent on laboratory evaluations of participants.

SUMMARY:
The purpose of this research study is to screen for metabolic abnormalities that are maternal risk factors for having a child with autism.

DETAILED DESCRIPTION:
The study will involve recruitment of 30 mothers of young children with ASD (ages 3-5 years) and 30 mothers of non-ASD children of similar age, respectively labelled ASD-moms and non-ASD-moms. In Phase 1, the levels of certain folate-related and oxidative stress biomarkers (folate, vitamin B12, vitamin E, homocysteine, methylmalonic acid, urinary isoprostanes) and MTHFR mutation analysis will be measured in all the mothers. The investigators expect that approximately 40-50% of the ASD-mothers and approximately 5-10% of the non-ASD-mothers will have abnormal homocysteine levels. In Phase 2, for those mothers with abnormal homocysteine levels, the investigators will treat them with a standard prenatal supplement for 4 weeks, and re-measure their biomarkers. The investigators expect 75-100% of the non-ASD mothers to respond, but only 25-50% of the ASD-mothers to respond. In Phase 3, for those mothers who did not respond to the standard prenatal supplement, the investigators will treat them with an optimized prenatal supplement for 4 weeks and remeasure their biomarkers. The investigators expect that 75-100% of the mothers of both groups will respond to this improved prenatal supplement.

ELIGIBILITY:
Mothers of children with autism (age 3-5) or typically-developing children (age 3-5) who are not currently taking prenatal vitamins/multivitamins.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Homocysteine level | 8-10 weeks
  Serial homocysteine level determination to assess response to supplementation with standard and optimized prenatal supplement in mothers exhibiting abnormal baseline homocysteine levels

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Woodruff, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James SJ, Melnyk S, Jernigan S, Pavliv O, Trusty T, Lehman S, Seidel L, Gaylor DW, Cleves MA. A functional polymorphism in the reduced folate carrier gene and DNA hypomethylation in mothers of children with autism. Am J Med Genet B Neuropsychiatr Genet. 2010 Sep;153B(6):1209-20. doi: 10.1002/ajmg.b.31094. PMID 20468076
- [Background] James SJ, Melnyk S, Jernigan S, Hubanks A, Rose S, Gaylor DW. Abnormal Transmethylation/transsulfuration Metabolism and DNA Hypomethylation Among Parents of Children with Autism. J Autism Dev Disord. 2008 Nov;38(10):1976. doi: 10.1007/s10803-008-0614-2. No abstract available. PMID 19011973
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials